CLINICAL TRIAL: NCT06812429
Title: Effects of Sodium-Glucose Co-transporter 2 Inhibitors on Inflammation
Acronym: EFSII
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Amanda Verma, Assistant Professor of Medicine, Principal Investigator, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202401169
Record Dates: First submitted 2025-02-01; First posted 2025-02-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Inflammation
Keywords: SGLT2 inhibitors; Dapagliflozin; Inflammation
MeSH Terms: conditions — Inflammation | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dapagliflozin group (Experimental): Participants in this arm receive dapagliflozin 10mg for three days.
  Interventions: Drug: Dapagliflozin (DAPA)

INTERVENTIONS:
Drug: Dapagliflozin (DAPA) — Participants will receive 10mg of Dapagliflozin per day for three days.

SUMMARY:
The research aims to understand how a specific type of medication called Sodium-glucose co-transporter 2 (SGLT2) inhibitors affect cardiorenal inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18
* Patient has no prior history or use of Sodium-Glucose Co-transporter 2 Inhibitors.
* Women who are surgically sterilized, amenorrheic for a year, on long-term contraceptives like intrauterine devices and implantable and injectable contraceptives.
* Willing and able to complete the outcome assessments.

Exclusion Criteria:

* History of cardiac diseases (Heart Failure, NSTEMI/STEMI, cardiomyopathies, myocarditis).
* Diagnosis of Type I Diabetes Mellitus.
* Symptomatic hypotension (symptoms of hypotension + Systolic blood pressure < 90).
* Estimated glomerular filtration rate <25 mL/minute/1.73 m2, with renal function test done within a year from the study enrollment date.
* Alcohol use disorder as defined by the NIAAA or use of controlled substances or smoking cigarettes.
* History of dapagliflozin or other Sodium-Glucose Co-transporter 2 Inhibitor sensitivity.
* Other concomitant disease or condition that the investigator deems unsuitable for the study, including psychiatric, behavioral, or cognitive disorders, sufficient to interfere with the patient's ability to understand and comply with the study instructions or follow-up procedures.
* Women who are pregnant or intend to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-04-05 (Actual); Study Completion 2025-04-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the markers of Inflammation at three days | From enrollment to the end of treatment at 3 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] USE OF SGLT2 INHIBITORS IN THE MANAGEMENT OF PATIENTS WITH HEART FAILURE POCKET GUIDE.
- [Background] Bonnet F, Scheen AJ. Effects of SGLT2 inhibitors on systemic and tissue low-grade inflammation: The potential contribution to diabetes complications and cardiovascular disease. Diabetes Metab. 2018 Dec;44(6):457-464. doi: 10.1016/j.diabet.2018.09.005. Epub 2018 Sep 26. PMID 30266577
- [Background] Cardiac And Kidney Benefits Of Dapagliflozin Are Associated With ApoM Levels In Patients With Heart Failure With Reduced Ejection Fraction
- [Background] Cowie MR, Fisher M. SGLT2 inhibitors: mechanisms of cardiovascular benefit beyond glycaemic control. Nat Rev Cardiol. 2020 Dec;17(12):761-772. doi: 10.1038/s41569-020-0406-8. Epub 2020 Jul 14. PMID 32665641
- [Background] Chirinos JA, Zhao L, Jia Y, Frej C, Adamo L, Mann D, Shewale SV, Millar JS, Rader DJ, French B, Brandimarto J, Margulies KB, Parks JS, Wang Z, Seiffert DA, Fang J, Sweitzer N, Chistoffersen C, Dahlback B, Car BD, Gordon DA, Cappola TP, Javaheri A. Reduced Apolipoprotein M and Adverse Outcomes Across the Spectrum of Human Heart Failure. Circulation. 2020 May 5;141(18):1463-1476. doi: 10.1161/CIRCULATIONAHA.119.045323. Epub 2020 Apr 2. PMID 32237898